CLINICAL TRIAL: NCT05631938
Title: A Phase I, Open-Label Study to Evaluate the Effect of Renal Impairment and Dialysis Treatment on the Pharmacokinetics of a Single 3 mg Cytisinicline Dose.
Brief Title: Study to Evaluate the Effect of Renal Impairment and Dialysis Treatment on the Pharmacokinetics of a Single 3 mg Cytisinicline Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-05
Record Dates: First submitted 2022-10-18; First posted 2022-11-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2023-10

CONDITIONS: Renal Impairment
Keywords: Dialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1: Normal Renal Function (Experimental): Participants with normal renal function receive a 3 mg single dose of cytisinicline.
  Interventions: Drug: cytisinicline
- Group 2: Mild Renal Impairment (Experimental): Participants with mild renal impairment receive a 3 mg single dose of cytisinicline.
  Interventions: Drug: cytisinicline
- Group 3: Moderate Renal Impairment (Experimental): Participants with moderate renal impairment receive a 3 mg single dose of cytisinicline.
  Interventions: Drug: cytisinicline
- Group 4: Severe Renal Impairment (Experimental): Participants with severe renal impairment receive a 3 mg single dose of cytisinicline.
  Interventions: Drug: cytisinicline
- Group 5: ESRD Participants Undergoing Dialysis (Experimental): Participants with ESRD undergoing dialysis receive a 3 mg single dose of cytisinicline on 2 occasions: after and prior to a dialysis session.
  Interventions: Drug: cytisinicline

INTERVENTIONS:
Drug: cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: cytisine

SUMMARY:
The primary objectives of this study are:

1. To obtain information on the pharmacokinetics of cytisinicline following a single oral dose in subjects with varying degrees of renal impairment relative to matched controls with normal renal function.
2. To investigate the extent of cytisinicline removal by hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Free written informed consent prior to any procedure required by the study.
* Ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the requirements of the study.
* Willingness to accept and comply with all study procedures and restrictions.
* Male or female subject between 18 and 75 years, inclusive, at Screening.
* Body mass index (BMI) of 18.0 to 35.0 kg/m^2, inclusive, at Screening.
* A female subject is eligible if she meets one of the following criteria:

  1. is of non-childbearing potential (underwent a permanent sterilization method [e.g., hysterectomy, bilateral salpingectomy and bilateral oophorectomy], is clinically diagnosed infertile, or is in a post-menopausal state); or
  2. is of childbearing potential and agrees to use an accepted contraceptive method from at least 28 days prior to dose administration (prior to first dose administration for Group 5) until at least 1 month after the end of study (EOS).
* Negative test results for anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), hepatitis B surface antigen (HBsAg) and anti-hepatitis C virus antibodies (anti-HCVAb).
* Stable concomitant medications for at least 7 days prior to dose administration (first dose administration for Group 5) and up to the EOS.

Additional Inclusion Criteria for Subjects with Renal Impairment (Groups 2 to 5)

* eGFR at Screening, determined by the Cockcroft-Gault equation, within:

  * 60-89 mL/min for Group 2 (mild renal impairment subjects).
  * 30-59 mL/min for Group 3 (moderate renal impairment subjects).
  * 15-29 mL/min for Group 4 (severe renal impairment subjects).
  * <15 mL/min for Group 5 (ESRD subjects)
* Subjects with ESRD are on dialysis for at least 3 months prior to Screening.
* Systolic blood pressure (SBP) 100-180mmHg, diastolic blood pressure (DBP) 50-105 mmHg, and pulse rate 50-100 bpm (inclusive), at Screening and Admission.

Additional Inclusion Criteria for Subjects with Normal Renal Function (Group 1)

* Estimated glomerular filtration rate (eGFR) ≥90 mL/min at Screening, determined by the Cockcroft-Gault equation.
* No clinically relevant abnormalities on clinical laboratory tests at Screening.
* Blood pressure and pulse rate at Screening within the following ranges:

  * SBP 90-140 mmHg, DBP 60-90 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects <65 years of age.
  * SBP 95-160mmHg, DBP 65-95 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects ≥65 years of age.

Exclusion Criteria:

* Known hypersensitivity/allergy reaction to cytisinicline substance or any of the excipients.
* History of renal, heart, and/or liver transplant.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere in a relevant manner with the absorption, distribution, metabolism, or excretion of the study treatment except for renal disease.
* Symptoms of an acute clinically relevant infection in the 4-week period preceding Screening (e.g., bacterial, viral, or fungal infection).
* History or clinical evidence of alcohol use disorder or substance use disorder according to Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) classification, within the 3-year period prior to Screening.
* Clinically relevant abnormalities on a 12-lead electrocardiogram (ECG), recorded after 5 min in the supine position at Screening.
* Currently using any creatine supplement.
* Nicotine consumption (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) from 48 hours prior to Admission.
* Excessive caffeine consumption, defined as ≥800 mg per day at Screening.
* Positive result in drugs-of-abuse or ethanol tests at Screening or Admission. NOTE: Subjects receiving stable treatment of methadone and benzodiazepines will be allowed to be enrolled in the study even if the urine drug screen test is positive.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
* Participation in any clinical trial within the previous 2 months.
* Loss of 250 mL or more blood within 3 months prior to screening.
* If female, positive pregnancy test in serum at Screening or positive pregnancy test in urine at Admission.
* If female, she is breast-feeding.

Additional Exclusion Criteria for subjects with Renal Impairment (Group 2 to 5)

* Presence of severe cardiac disease.
* History of severe renal artery stenosis.
* Presence of unstable diabetes mellitus.
* Acute, ongoing, recurrent, or chronic systemic disease other than renal function impairment that could interfere with the evaluation of the study results.
* Presence of any organ disorder, except for renal function impairment, which might interfere with the PK of cytisinicline.
* Use of any medication which might interfere with the PK of cytisinicline.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis), except for those related to renal impairment, at Screening.

Additional Exclusion Criteria for Subjects with ESRD (Group 5)

* Blood hemoglobin <10 g/dL at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetic (PK) Parameter: Maximum Observed Plasma Concentration (Cmax) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Time of Occurrence of Cmax (Tmax) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time of Dosing (t=0h) to the Time of the Last Measurable Concentration (AUC0-t) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Total AUC Extrapolated to Infinity (AUC0-∞) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Apparent Terminal Elimination Rate Constant (λz) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Apparent Terminal Elimination Half-Life (t1/2) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Fraction Unbound (fu) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Apparent Clearance (CL/F) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Plasma PK Parameter: Apparent Volume of Distribution (V/F) | pre-dose; 00:20, 00:40, 01:00, 01:20, 01:40, 02:00, 02:30, 03:00, 04:30, 06:00, 08:00, 12:00; 24:00, 36:00 and 48:00 hours:minutes post-dose
Urine PK Parameter: Amount of Drug Excreted in Urine (Ae) | pre-dose, 00:00-04:00 (groups 1-4), 00:00-06:00 (group 5), 04:00-08:00 (groups 1-4), 06:00-08:00 (group 5), 08:00-12:00, 12:00-24:00, 24:00-36:00 and 36:00-48:00 hours:minutes post-dose
Urine PK Parameter: Fraction of Unchanged Drug Excreted in Urine (fe) | pre-dose, 00:00-04:00 (groups 1-4), 00:00-06:00 (group 5), 04:00-08:00 (groups 1-4), 06:00-08:00 (group 5), 08:00-12:00, 12:00-24:00, 24:00-36:00 and 36:00-48:00 hours:minutes post-dose
Urine PK Parameter: Area Under the Urine Excretion Rate Curve From Time Zero to Last Measurable Observed Excretion Rate (AURC) | pre-dose, 00:00-04:00 (groups 1-4), 00:00-06:00 (group 5), 04:00-08:00 (groups 1-4), 06:00-08:00 (group 5), 08:00-12:00, 12:00-24:00, 24:00-36:00 and 36:00-48:00 hours:minutes post-dose
Urine PK Parameter: Renal Clearance (CLR) | pre-dose, 00:00-04:00 (groups 1-4), 00:00-06:00 (group 5), 04:00-08:00 (groups 1-4), 06:00-08:00 (group 5), 08:00-12:00, 12:00-24:00, 24:00-36:00 and 36:00-48:00 hours:minutes post-dose
Urine PK Parameter: Apparent Nonrenal Clearance (CLNR/F) | pre-dose, 00:00-04:00 (groups 1-4), 00:00-06:00 (group 5), 04:00-08:00 (groups 1-4), 06:00-08:00 (group 5), 08:00-12:00, 12:00-24:00, 24:00-36:00 and 36:00-48:00 hours:minutes post-dose
PK Parameter in Dialysate, Group 5 (ESRD on-dialysis): Amount of Drug Recovered From Each Dialysate Collection (AD) | Day 1 pre-dialysis, post-dialysis (before the hemodialysis is stopped), and for 1 minute every hour during hemodialysis
PK Parameter in Dialysate, Group 5 (ESRD on-dialysis): Cumulative Amount of Drug Recovered From the Dialysate (AD, total) | Day 1 pre-dialysis, post-dialysis (before the hemodialysis is stopped), and for 1 minute every hour during hemodialysis
PK Parameter in Dialysate, Group 5 (ESRD on-dialysis): Partial Area Under the Curve Estimated From Predialyzer Samples Collected From Start of Dialysis (t0) to End of Dialysis (t1) (AUCt0-t1) | Day 1 pre-dialysis, post-dialysis (before the hemodialysis is stopped), and for 1 minute every hour during hemodialysis
PK Parameter in Dialysate, Group 5 (ESRD on-dialysis): Dialysis Clearance (CLD) | Day 1 pre-dialysis, post-dialysis (before the hemodialysis is stopped), and for 1 minute every hour during hemodialysis
PK Parameter in Dialysate, Group 5 (ESRD on-dialysis): Fraction of the Administered Dose That is Recovered in the Dialysate (Frem) | Day 1 pre-dialysis, post-dialysis (before the hemodialysis is stopped), and for 1 minute every hour during hemodialysis

SECONDARY OUTCOMES:
Number of Participants With Clinically Significant Changes from Baseline in Body Weight | Baseline (pre-dose), 48 hours post-dose
Number of Participants With Clinically Significant Changes from Baseline in Systolic and Diastolic Blood Pressure | Baseline (pre-dose), 2, 6, 24, 36 and 48 hours post-dose
Number of Participants With Clinically Significant Changes from Baseline in Pulse Rate | Baseline (pre-dose), 2, 6, 24, 36 and 48 hours post-dose
Number of Participants With Clinically Significant Changes from Baseline in Body Temperature | Baseline (pre-dose), 2, 6, 24, 36 and 48 hours post-dose
Number of Participants With Clinically Significant Changes from Baseline in Hematology Values | Baseline (pre-dose), 48 hours post-dose
  Hematology assessments include hemoglobin, red blood cell (RBC) count, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width, white cell count with differential (neutrophil, eosinophil, basophil, lymphocyte and monocyte), platelet count and mean platelet volume.
Number of Participants With Clinically Significant Changes from Baseline in Biochemistry Values | Baseline (pre-dose), 48 hours post-dose
  Biochemistry values include sodium, potassium, glucose, creatinine, estimated creatinine clearance, total, direct and indirect bilirubin, alkaline phosphatase (ALP), lactate dehydrogenase (LDH), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), creatine phosphokinase (CPK), total protein and albumin.
Number of Participants With Clinically Significant Changes from Baseline in Coagulation Values | Baseline (pre-dose), 48 hours post-dose
  Coagulation assessments include prothrombin rate, prothrombin time-international normalized ratio (INR) and activated partial thromboplastin time (aPTT).
Number of Participants With Clinically Significant Changes from Baseline in Urinalysis Values | Baseline (pre-dose), 48 hours post-dose
  Urinalysis assessments include pH, specific gravity, protein, hemoglobin, glucose, ketones, bilirubin, nitrites, urobilinogen, and microscopy (if urine is available).
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | Groups 1 to 4: approximately 25 days; Group 5: approximately 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Guimarães, MD, PhD, Principal Investigator — Blueclinical, Ltd.
Locations (6):
- Portugal (3):
  - Hospital de Braga, Centro Clínico Académico Braga, Associação, Braga, Braga District
  - BlueClinical Phase I, Porto, Porto District
  - Early Phase Clinical Trials Unit | CHVNG/E + BlueClinical, Vila Nova de Gaia, Porto District
- Spain (3):
  - Hospital Universitario de La Princessa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No